CLINICAL TRIAL: NCT00293995
Title: Minimal Access Repair of Contralateral Hernias (MARCH Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04SG07
Record Dates: First submitted 2006-02-17; First posted 2006-02-20 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Unilateral Inguinal Hernia

ARMS (2):
- Laparoscopic repair (Other): Laparoscopic repair, with closure of contralateral patent processus vaginalis
  Interventions: Procedure: Repair of unilateral inguinal hernia
- Open repair (Other): Open repair
  Interventions: Procedure: Repair of unilateral inguinal hernia

INTERVENTIONS:
Procedure: Repair of unilateral inguinal hernia

SUMMARY:
Repair of unilateral inguinal hernia in infants. Laparoscopic repair, with closure of contralateral patent processus vaginalis if present, versus open repair

ELIGIBILITY:
Inclusion Criteria:

* unilateral inguinal hernia

Exclusion Criteria:

-

Ages: 0 Years to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
development of metachronous contralateral inguinal hernia | Until end of follow-up

SECONDARY OUTCOMES:
development of recurrent hernia | Until end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Agostino Pierro, Principal Investigator — Great Ormond Street Hospital
Locations (5):
- United Kingdom (5):
  - Addenbrookes Hospital, Cambridge
  - Royal Hospital for Sick Children, Edinburgh
  - Chelsea and Westminster Hospital, London
  - Great Ormond Street Hospital, London
  - King's College Hospital, London